CLINICAL TRIAL: NCT05327426
Title: Evaluating the Safety, Reactogenicity, and Immunogenicity of Intradermal Fractional Dose IPV (fIPV) in Combination With the Novel Mucosal Adjuvant, dmLT
Brief Title: Intradermal Fractional Dose IPV (fIPV) in Combination With dmLT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Jessica Crothers, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00001070
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Poliomyelitis
Keywords: polio; dmLT; mucosal adjuvant; fecal shedding; mOPV Challenge; fractional dose IPV (fIPV); intradermal vaccination
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- fIPV-dmLT (Experimental): Intradermal administration of fIPV with the addition of 0.47ug dmLT
  Interventions: Biological: Intradermal fractional dose inactivated polio vaccine (fIPV) in combination with recombinant double mutant heat labile toxin, LT(R192G/L211A), (dmLT); Biological: Monovalent oral poliomyelitis vaccine (mOPV), Sabin strain
- fIPV (Active Comparator): Intradermal administration of fIPV alone.
  Interventions: Biological: Intradermal fractional dose inactivated polio vaccine (fIPV); Biological: Monovalent oral poliomyelitis vaccine (mOPV), Sabin strain

INTERVENTIONS:
Biological: Intradermal fractional dose inactivated polio vaccine (fIPV) in combination with recombinant double mutant heat labile toxin, LT(R192G/L211A), (dmLT) — Sanofi's licensed IPOL trivalent inactivated polio vaccine (NDC 49281-860-78) delivered at the dose-sparing fractional volume of 1/5 the full dose (0.1mL) admixed with 0.47µg of recombinant double mutant [LT(R192G/L211A)] Enterotoxigenic Escherichia coli heat labile toxin (dmLT) adjuvant.
  Arms: fIPV-dmLT
Biological: Intradermal fractional dose inactivated polio vaccine (fIPV) — Sanofi's licensed IPOL trivalent inactivated polio vaccine (NDC 49281-860-78) delivered at the dose-sparing fractional volume of 1/5 the full dose (0.1mL).
  Arms: fIPV
Biological: Monovalent oral poliomyelitis vaccine (mOPV), Sabin strain — Monovalent oral polio vaccine (OPV) challenge administered as a test of mucosal immunity.

SUMMARY:
This is a single site, phase 1 study of dmLT as a mucosal adjuvant to control fecal viral shedding when used in combination with intradermally administered fractional dose trivalent IPV (fIPV). It will be a 2-arm, randomized, double-blind controlled trial of intradermal fIPV versus fIPV+dmLT in healthy adults with a monovalent oral polio vaccine (OPV) challenge administered as a test of mucosal immunity. A maximum of 30 healthy subjects will be recruited, all of whom will have received IPV only as part of their primary childhood immunization series (cohort 1); they will be randomized 2:1 to receive fIPV-dmLT or fIPV alone. A maximum of 27 participants will be recruited from an earlier pilot study population exposed to fIPV+/-dmLT and will provide follow-up samples for immunologic studies only (cohort 2).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 45 years old
2. Signed informed consent form prior to initiation of any study activity
3. Good general health as determined by review of medical history, physical exam, and basic laboratory screening
4. Agrees to complete all study visits and procedures
5. History of receipt of childhood polio vaccine series consisting of at least 3 doses of Inactivated Polio Vaccine (IPV). No history of receipt of OPV.
6. Neutralizing antibody titers > 1:8 for polio type 1

Exclusion Criteria:

* 1. Any condition (medical, psychiatric or behavioral) that, in the opinion of the investigator, would increase the volunteer's health risks in study participation or would increase the risk of not achieving the study's objectives (e.g., would compromise adherence to protocol requirements or interfere with planned safety and immunogenicity assessments) 2. Females of childbearing* potential only: currently lactating, breastfeeding, pregnant, or not agreeing to have repeated pregnancy tests prior to any study or challenge vaccination, and/or not having practiced adequate contraception** for 30 days prior to first study vaccination and/or not willing to continue using adequate contraception consistently for at least 90 days after the last study or challenge vaccination

  a. *Females can be considered not of childbearing potential if they are with current bilateral tubal ligation or occlusion, or post-hysterectomy, or post-bilateral ovariectomy, or post-menopause b. ** Adequate contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label, for example: i. Abstinence from penile-vaginal intercourse ii. Combined estrogen and progesterone oral contraceptives iii. Injectable progestogen iv. Implants of etonogestrel or levonorgestrel v. Contraceptive vaginal ring vi. Percutaneous contraceptive patches vii. Intrauterine device or intrauterine system viii. Male condom combined with a vaginal spermicide (foam, gel, film, cream or suppository), and/or progesterone alone oral contraceptive

  3. Symptoms of an acute self-limited illness, such as an upper respiratory infection, febrile illness (≥38.0°C (100.4°F), or gastroenteritis within 3 days of administration of IP including an oral temperature 4. History of antimicrobial treatment in the 10 days before administration of IP 5. History of a severe allergic reaction or anaphylaxis 6. Receipt of a vaccine within 21 days prior to the Investigational vaccination or anticipated receipt of any vaccine during the 28 days following Investigational vaccination 7. Receipt of a vaccine within the 21 days prior to OPV Challenge vaccination or anticipated receipt of any vaccine during the 28 days following OPV Challenge vaccination 8. Anticipated receipt of any investigational agent in the 28 days before or after receipt of investigational product without permission from the sponsor.

  9. Known history of hypersensitivity to any component of IPV or OPV to include: 2phenoxyethanol, formaldehyde, neomycin, streptomycin, polymyxin B erythromycin, and kanamycin 10. Receipt of polio vaccine within 12 months before the start of the study 11. Agrees not to and has no plans to travel outside the United States (US) until confirmation of cessation of vaccine virus shedding in stool 12. Having Crohn's disease or ulcerative colitis or having had major surgery of the gastrointestinal tract involving significant loss or resection of the bowel 13. Receipt of transfusion of any blood product or application of immunoglobulins within the 12 weeks prior to the first administration of study vaccine or planned use during the study period 14. Self-reported or suspected immunodeficiency, or receipt of immunosuppressive therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (inhaled, topical and intra-articular and epidural injections are allowed at this discretion of the investigator.

  15. Will have household or close professional contact during the mOPV challenge phase (C+0-C+28) of the study with individuals expected to be immunosuppressed (due to underlying condition or treatments) or individuals who have not yet completed their primary infant polio immunization series (i.e., three doses) 16. Will have household or close professional contact during the mOPV challenge phase (C+0-C+28) of the study with infants less than 6 months of age (e.g. neonatal nurses) or with pregnant women 17. Will have professional handling of food, catering or food production activities during the during the mOPV challenge phase (C+0-C+28) of the study 18. Indications of drug abuse or excessive use of alcohol that in the opinion of the investigator may interfere with their ability to comply with study related activities.

  19. Abnormal routine bowel habits as defined by fewer than three stools per week in the past 6 months 20. Regular use (weekly or more often) of laxatives, anti-diarrheal, or anti-constipation medications.

  21. Hepatitis B or C virus infection 22. Any confirmed or suspected immunosuppressive or immunodeficiency condition (human immunodeficiency virus [HIV] infection, or total serum immunoglobulin A (IgA) level below the testing laboratory lower limit of normal).

  23. Any hematological# or chemistry** parameter that is out of range of normal and is considered clinically significant by the investigator
  1. #Complete blood cell count (hemoglobin, hematocrit, white blood cell [WBC] and platelet count)
  2. **Creatinine, ALT, total bilirubin

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
mucosal immunity to poliovirus | 4 months
  Stimulation of mucosal immunity to poliovirus via comparison of fecal shedding dynamics using longitudinal stool collections following mOPV1 challenge in fIPV-dmLT recipients versus fIPV only recipients.

SECONDARY OUTCOMES:
Safety and local reactogenicity: systemic and local injection site adverse reactions (ARs) | 1 month
  Frequency of systemic and local injection site adverse reactions (ARs) defined as vaccine-related adverse events (AEs), graded by severity, occurring within 28 days of dosing
Safety: serious adverse events | 1 month
  percentage of subjects with at least one vaccine-related serious adverse event (SAE) occurring within 28 days of dosing
Systemic Immunogenicity: poliovirus-specific serum neutralizing antibody responses | 1 month
  poliovirus-specific serum neutralizing antibody responses in fIPV-dmLT recipients versus fIPV only recipients.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica W Crothers, MD, Principal Investigator — UVM Vaccine Testing Center
Locations (1):
- University of Vermont Vaccine Testing Center at the Larner College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated data will be made available to other researchers.